CLINICAL TRIAL: NCT04647279
Title: Clinical Study of New MRI Sequences in Spine and Joint
Brief Title: New MRI Sequences in Spine and Joint
Acronym: NMSSJ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, ShaoLin Li, Director of Radiology Department, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY.FSK.004
Record Dates: First submitted 2020-11-27; First posted 2020-11-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Degeneration of Spine and Osteoarticular
Keywords: Magnetic resonance imaging; Low back pain; Disk degeneration; Ultrashort echo time; Osteoarticular degeneration
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal control group: Diagnostic Test: Quantitative MRI imaging IR-UTE, UTE-MT, Maigc, Ideal IQ, DTI, and IVIM
  Interventions: Diagnostic Test: Dual-emission X-ray Absorptiometry
- Osteopenia: Diagnostic Test: Quantitative MRI imaging IR-UTE, UTE-MT, Maigc, Ideal IQ, DTI, and IVIM
  Interventions: Diagnostic Test: Dual-emission X-ray Absorptiometry
- Osteoporosis: Diagnostic Test: Quantitative MRI imaging IR-UTE, UTE-MT, Maigc, Ideal IQ, DTI, and IVIM
  Interventions: Diagnostic Test: Dual-emission X-ray Absorptiometry

INTERVENTIONS:
Diagnostic Test: Dual-emission X-ray Absorptiometry — The recruiters were divided into osteoporosis, osteopenia and normal by dual emission X-ray absorptiometry.

SUMMARY:
Low back pain and osteoarticular degeneration or injury is the leading worldwide cause of years lost to disability, accounting for 17 % of all patients with disabilities and its burden is growing alongside the increasing and aging population. The anatomical regions of the intervertebral disc include the central nucleus pulposus, the peripheral fibrocartilaginous annulus fibrosus, and the superior and inferior cartilaginous endplates (CEP). The CEP is a thin layer of hyaline cartilage located between the avascular intervertebral disc and the bony vertebral endplate. The endplate cartilage consists of chondrocytes interspersed throughout an extracellular matrix of proteoglycans, collagen (types I and II), and water. It plays an important role in the function and homeostasis. The CEP has been considered the pathway between the largely avascular disk tissues and the blood supply of the vertebral body and thus provides nutrition for disk cells. Many musculoskeletal tissues, including the CEP, cartilage-bone interface of articular joints, entheses, tendons, and ligaments, have components with very short T2 values (much less than 1 msec), which are orders of magnitude shorter than that of the nucleus of the disk (~100 msec). In a conventional pulse sequence, such as proton density-weighted spin-echo (SE) or fast SE, with standard clinical section profile, the minimum echo time (TE) is typically 10 msec, which is much longer than that needed to capture the short-lived signal from these tissues. Recently, ultrashort echo sequence UTE technology has been introduced, and the TE time can be as low as 0.008ms. This range of TE is sufficient to capture signals from the cartilage endplate before it decays. With using new MRI technology, such as IR-UTE, UTE-MT, UTE-T2*mapping, Maigc, DTI, and IVIM, which can quantitative tissues that have previously been "invisible" at conventional MR imaging, and provide imaging basis for early diagnosis of injury at molecular level. The purpose of this study was to investigate the clinical application value of different MRI sequences in spine and joint.

ELIGIBILITY:
Inclusion Criteria:

* 1.The patient had history and clinical symptoms of low back pain and joint sports injury 2.The patient had a history of osteoporosis; 3.There was no contraindication of MRI; 4.The patient who has clear lumbar intervertebral disc degeneration or herniation or osteoporosis or joint sports injury found by routine CT or MRI examination, and the clinical symptoms were consistent with the image.

Exclusion Criteria:

* 1. Patients with previous history of lumbar or joint surgery; 2. Patients with congenital bone deformity; 3. Patients with history of lumbar tumor and infection; 4. Cognitive function is limited or mental illness can not cooperate with imaging.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All suspected patients with osteoporosis and low back pain meet the inclusion criteria will include in this study. And patients who meet the criteria of the normal control group will include in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
New MRI sequences in the diagnosis of spine and joint | 2 years
  Quantitative MRI imaging(such as IR-UTE, UTE-MT, UTE-T2*mapping, Maigc, Ideal IQ, DTI, and IVIM) used to quantitative diagnosis of disk degeneration, osteoporosis, osteoarticular degeneration etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawakami M, Tamaki T, Hayashi N, Hashizume H, Nishi H. Possible mechanism of painful radiculopathy in lumbar disc herniation. Clin Orthop Relat Res. 1998 Jun;(351):241-51. PMID 9646768
- [Background] Bae WC, Statum S, Zhang Z, Yamaguchi T, Wolfson T, Gamst AC, Du J, Bydder GM, Masuda K, Chung CB. Morphology of the cartilaginous endplates in human intervertebral disks with ultrashort echo time MR imaging. Radiology. 2013 Feb;266(2):564-74. doi: 10.1148/radiol.12121181. Epub 2012 Nov 28. PMID 23192776
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Lotz JC, Fields AJ, Liebenberg EC. The role of the vertebral end plate in low back pain. Global Spine J. 2013 Jun;3(3):153-64. doi: 10.1055/s-0033-1347298. Epub 2013 May 23. PMID 24436866
- [Background] Gatehouse PD, Bydder GM. Magnetic resonance imaging of short T2 components in tissue. Clin Radiol. 2003 Jan;58(1):1-19. doi: 10.1053/crad.2003.1157. PMID 12565203
- [Background] Bae WC, Dwek JR, Znamirowski R, Statum SM, Hermida JC, D'Lima DD, Sah RL, Du J, Chung CB. Ultrashort echo time MR imaging of osteochondral junction of the knee at 3 T: identification of anatomic structures contributing to signal intensity. Radiology. 2010 Mar;254(3):837-45. doi: 10.1148/radiol.09081743. PMID 20177096
- [Background] Bae WC, Du J, Bydder GM, Chung CB. Conventional and ultrashort time-to-echo magnetic resonance imaging of articular cartilage, meniscus, and intervertebral disk. Top Magn Reson Imaging. 2010 Oct;21(5):275-89. doi: 10.1097/RMR.0b013e31823ccebc. PMID 22129641
- [Background] Pfirrmann CW, Metzdorf A, Zanetti M, Hodler J, Boos N. Magnetic resonance classification of lumbar intervertebral disc degeneration. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1873-8. doi: 10.1097/00007632-200109010-00011. PMID 11568697
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424